CLINICAL TRIAL: NCT05683041
Title: Prevention of Intra-uterine Adhesions Following Laparoscopic and Laparotomic Myomectomy
Acronym: PALLM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ONZ-2022-0355
Record Dates: First submitted 2022-12-20; First posted 2023-01-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Myoma
Keywords: Postoperative adhesions; Intrauterine adhesions; Myomectomy; Laparoscopic myomectomy; Laparotomic myomectomy; Adhesion prevention; Antiadhesion method
MeSH Terms: conditions — Myoma; Gynatresia

STUDY DESIGN:
Intervention Model Description: This study investigates whether the use of an intrauterine gel can prevent the development of these adhesions. The application of antiadhesion gel is compared to no gel.
Who Masked: Participant, Care Provider, Investigator
Masking Description: None of the participants will be informed of the allocated treatment by the surgeon or the personnel present in the OR. The medical record will not reveal any information whether antiadhesion gel was applied at the end of the procedure. In the case that the surgeon is the same person as the gynaecologist doing the second-look hysteroscopy, blinding is assured by notification of treatment allocation if the surgeon has left the operating room.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intrauterine gel application (Experimental): Application of Hyalobarrier intrauterine after myomectomy.
  Interventions: Device: Hyalobarrier
- no intra-uterine gel application (No Intervention): No application of Halobarrier intrauterine after myomectomy.

INTERVENTIONS:
Device: Hyalobarrier — Hyalobarrier is a viscous, transparent gel and is used as a preventive measure for post-operative adhesions in the abdominal and uterine cavity.
  Other Names: anti-adhesive gel
  Arms: intrauterine gel application

SUMMARY:
Clinical study on the prevention of intrauterine adhesions after laparoscopic or laparotomic myomectomy.

Myomas are common in women of reproductive age and myomectomy can lead to intra-uterine adhesions, which can be detrimental to fertility. This study investigates whether the use of an intrauterine gel can prevent the development of these adhesions.

DETAILED DESCRIPTION:
Design:

Double-blind, randomized controlled pilot trial.

Participant:

* age between 18 and 45 years.
* intramurale and/or subserosal myoma (FIGO 3-6), and/or hybrid myoma (with a connection to the endometrium and serosa (FIGO 2-5), who are scheduled for laparoscopic / laparotomic myomectomy.
* absence of intra-uterine adhesions on preoperative diagnostic hysteroscopy

Treatment:

Application of intrauterine Hyalobarrier® gel endo at time of surgery

Control:

No application of Hyalobarrier® gel endo

Follow up:

Second-look hysteroscopy after 3months

To blind all trial participants and gynaecologists doing second-look hysteroscopy, 10 ml of a sterile ultrasound gel will be applied into the vagina at the end of the procedure in all women regardless of their treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 45 years.
* intramurale and/or subserosal myoma (FIGO 3-6), and/or hybrid myoma (with a connection to the endometrium and serosa (FIGO 2-5), who are scheduled for laparoscopic / laparotomic myomectomy.
* absence of intra-uterine adhesions on preoperative diagnostic hysteroscopy

Exclusion Criteria:

* pregnancy.
* laparoscopic or laparotomic myomectomy in combination with an operative hysteroscopy.
* presence of endometritis.
* other antiadhesion methods

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only woman included with uterus.
Enrollment: 30 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Adhesion formation postoperatief. | 3 months post surgery
  The presence of intra-uterine adhesions on a second look hysteroscopy.

SECONDARY OUTCOMES:
Severity of adhesion formation | 3 months post surgery, at the time of the hysteroscopy.
  American Fertility Society classification (AFS) and classification of Valle and Sciarra are used to describe the severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No